CLINICAL TRIAL: NCT05330884
Title: Efficacy of BCG Revaccination Compared With Oral Chemoprophylaxis in Household Contacts Aged 6-18 Years for Prevention of Tuberculosis Disease - A Phase III Open Labelled Randomised Controlled Trial
Brief Title: BCG Revaccination in Children and Adolescents
Acronym: BRiC
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: changes in protocol
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: Institute of Child Health, Chennai (Unknown); All India Institute of Medical Sciences (Other); The Grant Medical College & Sir J.J. Group of Hospitals (Other Government); All India Institute of Medical Sciences, Bhubaneswar (Other); Rajendra Institute of Medical Sciences, Ranchi (Unknown); National Institute of Tuberculosis and Respiratory Diseases, New Delhi (Unknown); Rajiv Gandhi Hospital, Chennai (Unknown); Madurai Medical College (Other); Government Vellore Medical College, Vellore (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022 005
Record Dates: First submitted 2022-03-28; First posted 2022-04-15 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Tuberculosis Infection; Tuberculosis
Keywords: BCG; Anti tuberculous Chemoprophylaxis; LTBI; TB; Vaccine
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis | interventions — BCG Vaccine; Chemoprevention

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomised trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vaccine - Bacille Calmette-Guérin vaccine (BCG ) (Experimental): Bacille Calmette-Guérin vaccine (BCG ) dose 0.1ml intradermal
  Interventions: Biological: BCG vaccine
- Chemoprophylaxis - as per NTEP guidelines (Other): Oral chemoprophylaxis: according to the existing standard of care (NTEP guidelines) Either six months of isoniazid (10mg/kg) or Rifapentine and isoniazid weekly for 3 months for DS TB Levofloxicillin or standard of care drug for DR TB: 15-20mg/kg/day
  Interventions: Drug: Oral Chemoprophylaxis

INTERVENTIONS:
Biological: BCG vaccine — 0.1ml BCg vaccine to be given intradermally
  Arms: vaccine - Bacille Calmette-Guérin vaccine (BCG )
Drug: Oral Chemoprophylaxis — Oral chemoprophylaxis will be standard of care - either 6 months of Isoniazid or 3 months of weekly Isoniazid and Rifapentine
  Arms: Chemoprophylaxis - as per NTEP guidelines

SUMMARY:
Bacille Calmette Guerin (BCG) vaccine is one of the most used vaccines of the world, to reduce the risks of natural tuberculous infection. The efficacy of BCG vaccination in newborns is well known and has a documented protective effect against meningitis and disseminated TB in children. However, there is considerable uncertainty on BCG revaccination. It is known that BCG revaccination enhances immune responses, but it is yet to be established if BCG revaccination can help prevent TB disease in household contacts.

The primary aim of this study is to assess the efficacy of BCG revaccination compared to oral chemoprophylaxis in preventing TB disease in house hold contacts aged 6-18 years.

The study is designed as a multicentre randomised controlled trial with two groups of healthy household contacts aged 6-18 years receiving either the BCG vaccine or oral chemoprophylaxis. They will be followed up for 24 months to compare the incidence of TB disease in each arm.

DETAILED DESCRIPTION:
Objectives

Primary:

To demonstrate the effect of BCG revaccination in comparison to oral chemoprophylaxis on the incidence of Mycobacterium tuberculosis disease in healthy household contacts aged 6-18 years.

Secondary:

* To compare the safety of BCG revaccination with oral chemoprophylaxis
* To study the efficacy of BCG revaccination in comparison to oral chemoprophylaxis in preventing Mycobacterium tuberculosis infection
* To study the immunogenicity of BCG revaccination

Methodology The aim of this study is to assess the efficacy of BCG revaccination compared to oral chemoprophylaxis in preventing TB disease in house hold contacts aged 6-18 years. The study is designed as a multicentre randomised controlled trial with two groups of healthy household contacts aged 6-18 years receiving either the BCG vaccine or oral chemoprophylaxis. A total of 9200 children will be recruited across 7 sites in India. Children will be randomised into 2 study arms: 1) BCG; 2) Oral chemoprophylaxis.

All children will be household contacts of microbiologically confirmed pulmonary TB patients. Contacts of MDR TB adults will also be included in the study. Both C-Tb skin test positive and negative children will be included. Similarly, both well-nourished and malnourished children will be included. All children will be followed up for 24 months post recruitment and the incidence of TB (all forms - PTB / EPTB) will be compared between the groups. TB will be diagnosed as per the NTEP guidelines and LTBI will be based on the C-TB skin test results.

Immunology bloods will be done in 10% of the participants - 920 children at baseline, 3, 6 12 and 24 months. The immunology component of this trial is designed so as to decipher clearly the effects of BCG revaccination on adaptive and innate cell responses. Full Blood Count for Monocyte/Lymphocyte ratio, Whole Blood culture for Intracellular Staining, Innate assays, Mycobacterial Growth Inhibition Assay and acute phase proteins will be performed between groups

ELIGIBILITY:
Inclusion Criteria:

* Healthy household contacts aged 6 to 18 yr
* Previously vaccinated with BCG at birth or least 5 years ago - evidence of scar or documented immunisation record.
* General good health - through history and baseline screening
* Agrees to continue in the study for 2 years post enrollment
* Children previously treated for LTBI and completed treatment at least 6 months ago - can also be included. However, they should be current HHC

Exclusion Criteria:

* Any acute illness on recruitment day (Evaluate the child again at a later stage)
* Fever ≥38 degree Celsius on recruitment day (Evaluate the child again at a later)
* History of autoimmune disease
* Pregnancy - female participants > 15 years of age will have pregnancy test done after caretakers and participants informed consent
* Evidence of active TB disease
* On treatment for active TB disease or LTBI
* HIV positive or any history or present possible immunodeficiency condition
* History of allergic reactions to vaccines in past
* Pre-existing liver dysfunction
* ALT/AST is ≥ 3 times upper limit of normal (ULN) in the presence of symptoms or ≥ 5 times the ULN in the absence of symptoms and/or total bilirubin greater than ULN along with raised ALT/AST.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 9200 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of TB (all forms - PTB / EPTB) as per NTEP guidelines | over 24 months
  Incidence of TB in BCG revaccinated and oral chemoprophylaxis groups (age and gender stratified)

SECONDARY OUTCOMES:
Adverse events | 24 months
  Incidence of adverse events in children in each arm
MTB infection | 24 months
  Incidence of MTB infection in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Aishwarya Venkataraman, MRCPCH, Principal Investigator — ICMR-National Institute for Research in Tuberculosis
Locations (1):
- Dr Aishwarya Venkataraman, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Undecided